CLINICAL TRIAL: NCT05264428
Title: The Effect of Honey on Lessening the Withdrawal Symptoms According to the Body Constitution
Brief Title: The Effect of Honey on Lessening the Withdrawal Symptoms
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Buddhist Tzu Chi General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P00001592
Record Dates: First submitted 2022-02-11; First posted 2022-03-03 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-02

CONDITIONS: Smoking Cessation; Withdrawal Symptoms
MeSH Terms: conditions — Smoking Cessation; Substance Withdrawal Syndrome | interventions — Honey; Water

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Participants need to drink honey every day for four weeks.
  Interventions: Dietary Supplement: Honey
- Control group (Placebo Comparator): Participants need to drink water every day for four weeks.
  Interventions: Dietary Supplement: Water

INTERVENTIONS:
Dietary Supplement: Honey — Participants need to drink honey every day for four weeks.
  Arms: Experimental group
Dietary Supplement: Water — Participants need to drink water every day for four weeks.
  Arms: Control group

SUMMARY:
This project investigates the effect of honey on lessening the withdrawal symptoms according to the body constitution.

ELIGIBILITY:
Inclusion Criteria:

* the cessation clinic patients aged more than 18
* only take Champix for smoking cessation

Exclusion Criteria:

* diabetes, cancer, renal disease
* with wet and hot body constitution
* allergic to honey
* accepting traditional Chinese medicine intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-09-03 (Actual); Primary Completion 2023-02-28 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Fagerstrom Test for Nicotine Dependence | Before and after the 4-week trial, 3 and 6 months after the trial
  Change from baseline Fagerstrom Test for Nicotine Dependence at 4 weeks, 3 and 6 months after the trial. Fagerstrom Test for Nicotine Dependence is ranged from 0-10. The higher score the higher dependence on Nicotine.
Minnesota Nicotine Withdrawal Scale | Before and after the 4-week trial
  Change from baseline Minnesota Nicotine Withdrawal Scale at 4 weeks. The Minnesota Nicotine Withdrawal Scale is ranged from 0-84. The higher score indicates more severe withdrawal syndromes.

SECONDARY OUTCOMES:
Body Constitution Questionnaire | Before and after the 4-week trial
  Change from baseline Body Constitution Questionnaire at 4 weeks. The Body Constitution Questionnaire contains 9 sub-scales, each is ranged from 0-100. The higher score indicates the likelihood of the body constitution.
Tobacco Craving Questionnaire | Before and after the 4-week trial
  Change from baseline Tobacco Craving Questionnaire at 4 weeks. The Tobacco Craving Questionnaire contains 47 items that ranged from 1-7. The higher score indicates the higher craving for tobacco.
Depression Anxiety Stress Scales-21 | Before and after the 4-week trial
  Change from baseline Depression Anxiety Stress Scales-21 at 4 weeks. The Depression Anxiety Stress Scales-21 contains 3 sub-scales, each is scored form 0-28. The higher score indicates the more negative condition.
WHOQOL-BREF | Before and after the 4-week trial
  Change from baseline WHOQOL-BREF at 4 weeks. WHOQOL-BREF contains 4 domains, each domain will be calculated to a score ranged from 0-100. The score of 100 indicates satisfaction of QOL.
Pittsburgh sleep quality index | Before and after the 4-week trial
  Change from baseline Pittsburgh sleep quality index at 4 weeks. The Pittsburgh sleep quality index ranged from 0 to 21. The higher score indicates more severe difficulties in sleep.
Readiness to Quit Ladder | Before and after the 4-week trial
  Change from baseline Readiness to Quit Ladder at 4 weeks. The Readiness to Quit Ladder is rated from 1 to 10. The higher score indicated better readiness to quit smoking.

CONTACTS AND LOCATIONS:
Locations (1):
- Hualien Tzu Chi Hospital, Hualien City, Taiwan